CLINICAL TRIAL: NCT00891956
Title: The Role of Family Functioning in Adaptation to Being a Caregiver of an Individual With Rett Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909132; 09-HG-N132
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2016-01-13

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Rett syndrome (RS) is a panethnic (affecting all ethnicities) neurodevelopmental (impairment of the growth and development of the brain) disorder affecting primarily females. RS is characterized by the loss of intellectual functioning, fine and gross motor skills, and communicative abilities after a period of seemingly normal development.
* Caregivers of individuals with RS face many psychosocial challenges. The stressors can be grouped into the following six categories: emotional difficulties, health-related stressors, uncertainty about their daughter s illness, rejection by their social environment, lack of available or competent experts, and unfavorable comparison with healthy children.
* Researchers are making a significant contribution to the adaptation literature with a focus on family functioning and to the little psychosocial research that exists on families with RS.
* Researchers hope to narrow down the most important areas on which to focus for intervention strategies in families with RS.

Objectives:

* To describe family functioning, perceived illness burden, self-efficacy, types of coping methods, and adaptation in caregivers of individuals with RS to examine the relationships between these variables and the outcomes of family functioning and adaptation.
* To examine the extent to which appraisals of being a caregiver of an individual with RS and methods of coping are associated with family functioning.
* To examine the extent to which appraisals of being a caregiver of an individual with RS, methods of coping, and family functioning are associated with caregiver adaptation.

Eligibility:

- Eligibility is based on answering yes to the following three questions: Are you 18 years old or older? Are you the caregiver of a child diagnosed with Rett Syndrome? and Does the child with Rett Syndrome currently reside in your home with you?

Design:

* Participants in this cross-sectional research design will answer a quantitative survey that includes some open-ended questions. The cross-sectional study involves a one-time self-administered questionnaire that takes approximately 20 to 30 minutes to complete.
* The survey will be available in paper and electronic versions and includes demographics questions, measures of perceived illness burden, parental self-efficacy, coping methods, family functioning, and adaptation. Participants also will answer open-ended questions related to the individual s diagnosis.
* Participants may withdraw from the study at any point up until submission of the survey and may skip any question.
* Participants who experience psychological distress as a result of taking the survey are advised to contact the researcher. Study coordinators at the various clinics from which participants will be recruited will be notified of the possibility of adverse events and instructed to direct any members who experience distress to the appropriate professional services.
* Participants will receive a small financial compensation for completing the survey.

DETAILED DESCRIPTION:
This study aims to investigate the predictors of family functioning and adaptation in caregivers of individuals with Rett Syndrome (RS), a neurodevelopmental disorder affecting primarily females. After an apparently normal prenatal and postnatal period of development, individuals with RS lose intellectual functioning, fine and gross motor skills including purposeful hand use, and communicative abilities. Individuals with RS also experience a host of other medical problems including seizures and respiratory dysfunction. Prior research demonstrates that caregivers of individuals with RS experience more stress than normative samples and that family functioning plays a role in maternal mental health. However, there is much that is not understood about how cognitive appraisals (thoughts that assess the circumstances), coping methods, and family functioning are related to caregiver adaptation in this population. This study is based on Thompson and colleagues Transactional Stress and Coping Model which conceptualizes family functioning and adaptation to being a caregiver of an individual with RS. A cross-sectional research design using quantitative methodology will explore the relationships between perceived illness burden, self-efficacy, coping methods, family functioning and adaptation. In addition, an open-ended section will be included to qualitatively describe the role of family relationships on the caregivers perception of their ability to care for their child with RS. Caregivers of individuals with RS will be recruited through an international RS organization, a national RS educational meeting, and several national RS clinics. Eligible participants will be able to complete a paper or online version of the survey.

ELIGIBILITY:
* INCLUSION CRITERIA:
* The study population will consist of men and women ages 18 or older who are the primary caregivers of a child with Rett Syndrome.
* The parent may be a biological or adoptive parent or other primary caregiver and the child must reside with the primary caregiver.
* Individuals of all ethnic, religious, socioeconomic, and educational backgrounds and from a variety of geographic locations in the United States will be included.

EXCLUSION CRITERIA:

-Participants must be able to read and write in English, as it is essential for the researchers to be able to understand participants responses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2009-04-24; Study Completion 2016-01-13

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Hagberg B. Rett syndrome: clinical peculiarities and biological mysteries. Acta Paediatr. 1995 Sep;84(9):971-6. doi: 10.1111/j.1651-2227.1995.tb13809.x. PMID 8652969
- [Background] Lotan M, Ben-Zeev B. Rett syndrome. A review with emphasis on clinical characteristics and intervention. ScientificWorldJournal. 2006 Dec 6;6:1517-41. doi: 10.1100/tsw.2006.249. PMID 17160339
- [Background] Weaving LS, Ellaway CJ, Gecz J, Christodoulou J. Rett syndrome: clinical review and genetic update. J Med Genet. 2005 Jan;42(1):1-7. doi: 10.1136/jmg.2004.027730. PMID 15635068